CLINICAL TRIAL: NCT06423339
Title: A Comparative Study Between Ultrasound Guided Genicular Nerve Block Combined With Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee Block Versus Adductor Canal Block in Total Knee Replacement
Brief Title: Comparison Between (GNB) Combined With (IPACK) Block Versus ACB in TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAMSU R80/2024
Record Dates: First submitted 2024-04-27; First posted 2024-05-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive genicular nerve block combined with interspace between the popliteal artery and the capsule of the posterior knee block(IPACK)
  Interventions: Procedure: Ultrasound guided Genicular nerve block; Procedure: Interspace between the popliteal artery and the capsule of the popliteal artery and the capsule of the posterior knee; Drug: Bupivacaine Hydrochloride
- Group B (Experimental): Group B will receive ultrasound guided sub-sartorial Adductor canal block (ACB)
  Interventions: Procedure: Adductor canal block; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Procedure: Ultrasound guided Genicular nerve block — Ultrasound guided genicular nerve block
  Arms: Group A
Procedure: Interspace between the popliteal artery and the capsule of the popliteal artery and the capsule of the posterior knee — Ultrasound guided Interspace between the popliteal artery and the capsule of the popliteal artery and the capsule of the posterior knee
  Arms: Group A
Procedure: Adductor canal block — Ultrasound guided sub-sartorial Adductor canal block
  Arms: Group B
Drug: Bupivacaine Hydrochloride — Pupivacaine 0.5% in 20 ml vial
  Other Names: Sunnypivacaine

SUMMARY:
The patients will be randomized into 2 groups, named group A, B.

Group A: The patients will receive Ultrasound guided Genicular nerves block combined with Ultrasound guided IPACK block.

Group B: The patients will receive Adductor canal block which will be the control group.

The Numerical Rating Scale (NRS) will be used to assess pain intensity. Preoperatively, all study subjects will be trained to use NRS pain scores.

The spinal block will be performed.

In group A, 15 mL of bupivacaine 0.25% with 2.5 g/mL adrenaline at a concentration 1:4,00,000 will be administered immediately following skin closure. GNB will be performed by using the linear ultrasound probe (10-15 MHz) Sono site M-turbo ultrasonography to scan the long bone shaft with up and down movement to recognize the epicondyle of the tibia and femur. The junctions between the epicondyle and the shafts of the femur and tibia are where the genicular arteries are located; these junctions will be defined as the periosteal areas. The superior lateral, superior medial and inferior medial genicular arteries accompany each genicular nerve. After confirmation of the genicular artery by color Doppler, the needle will be introduced using the in-plane approach and presented in the long axis view. The target point of the needle insertion will be the needle tip beside a genicular artery. Then, a 5 mL volume will be administered after gentle aspiration to prevent a faulty intra-arterial injection at 3 target locations: the superior lateral, superior medial and inferior medial genicular nerves.

This will be Followed by the procedure for the IPACK block.

In group B, A 22 Gauge 80 mm needle will be guided from lateral to medial to this area called the adductor canal using in-plane technique. 20 mL of 0.5% bupivacaine will be injected with peri-arterial spread after negative aspiration under sterile conditions. TKA will be performed by an orthopedic surgeon by placing three-compartment prostheses with a minimally invasive mini-midvastus approach and using hand-mixed cementing techniques.

DETAILED DESCRIPTION:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B. An independent data manager of computer generated software will be responsible for randomization, assigning the patients to the groups using sequentially numbered, sealed, opaque envelopes containing computer generated random numbers, accessible only to the anesthesiologist performing the block. The subjects will be randomly allocated to one of the two groups.

Group A: The patients will receive Ultrasound guided Genicular nerves block combined with Ultrasound guided IPACK block.

Group B: The patients will receive Adductor canal block which will be the control group.

History taking, clinical examination and routine laboratory investigation will be performed preoperatively, and the patients will be instructed to fast for 8 hours preoperative for solids and 2 hours for clear fluids. On arrival to the operation room, intravenous access will be established and acetated ringer will be infused by rate 10ml/kg. ECG, noninvasive blood pressure and arterial oxygen saturation will be monitored routinely. The Numerical Rating Scale (NRS) will be used to assess pain intensity. Preoperatively, all study subjects will be trained to use NRS pain scores.

In the operating room, a peripheral 20 G intravenous (IV) cannula will be inserted. The baseline parameters of five lead electrocardiogram (ECG), non invasive blood pressure and peripheral oxygen saturation will be recorded. IV midazolam 0.02 mg/kg will be administered. The spinal block will be performed using either a 25 or 27 G spinal needle in the sitting position at the L3-L4 or L4-L5 intervertebral space with a 2.5-3 mL hyperbaric bupivacaine 0.5%. The sensory block (to cold and pinprick) to the 10th thoracic dermatome or above will be the target of the spinal block to start the surgery. Hypotension will be defined as ≥20% decrease in blood pressure from baseline measurements and managed by IV Ephedrine6 mg boluses.

In group A, 15 mL of bupivacaine 0.25% with 2.5 g/mL adrenaline at a concentration 1:4,00,000 will be administered immediately following skin closure. GNB will be performed by using the linear ultrasound probe (10-15 MHz) Sono site M-turbo ultrasonography to scan the long bone shaft with up and down movement to recognize the epicondyle of the tibia and femur. The junctions between the epicondyle and the shafts of the femur and tibia are where the genicular arteries are located; these junctions will be defined as the periosteal areas. The superior lateral, superior medial and inferior medial genicular arteries accompany each genicular nerve. After confirmation of the genicular artery by color Doppler, the needle will be introduced using the in plane approach and presented in the long axis view. The target point of the needle insertion will be the needle tip beside a genicular artery. Then, a 5 mL volume will be administered after gentle aspiration to prevent a faulty intra arterial injection at 3 target locations: the superior lateral, superior medial and inferior medial genicular nerves.

This will be Followed by the procedure for the IPACK block initiated by the visualization of the popliteal artery and posterior surface of the distal femur. Then, the image of the femoral condyles and the popliteal artery will be obtained. A 20G 22G 80 mm needle will be inserted in a medial to the lateral plane, parallel to the femur in the middle area between the popliteal artery and the femur. 20 mL of the local anesthetic solution will be given into this space in increments, ensuring the adequate and equal distribution of the anesthetic agent.

In group B, after placing the patients in the supine position, the linear probe of ultrasound (13-6 MHz) will be moved from cephalad to caudal and the superficial femoral artery will be visualized in the short axis, medial to the vastus medialis, lateral to the sartorius muscle, and anterior to the adductor magnus muscle.

A 22 Gauge 80 mm needle will be guided from lateral to medial to this area called the adductor canal using in-plane technique. 20 mL of 0.5% bupivacaine will be injected to with peri-arterial spread after negative aspiration under sterile conditions. TKA will be performed by an orthopedic surgeon by placing three-compartment prostheses with a minimally invasive mini-midvastus approach and using hand-mixed cementing techniques.

The outcome:

The primary outcome will be the total postoperative morphine consumption during the first two postoperative days. NRS will be assessed at 0, 6, 12, 24 and 48 h postoperatively. The period between the end of surgery and the first request for rescue analgesia (NRS >3) will be considered the time to the first request. Postoperative analgesia, IV paracetamol (1 g/6 h) and IV ketorolac (30 mg/12 h), will be administered to all patients. The pain will be assessed at rest and during movement using NRS (metric score 0-10 for pain severity assessment: mild pain = 1-3, moderate = 4-7 and severe = 8 and above) on the first and second days. When NRS will be >3, rescue analgesia (morphine 3 mg IV) will be given and repeated whenever required.

The secondary outcome will be assessment of Postoperative functional outcomes and knee rehabilitation parameters including quadriceps motor strength score measured by straight leg raising (SLR), knee range of motion (ROM) and time up and go (TUG) test. SLR will be assessed on a scale ranging from 0 to 5 as follows: 0 = unable to contract muscles, 1 = muscles twitch, the limb does not move, 2 = able to move the limb with gravity elimination and passive assistance, 3 = able to move the limb against gravity without resistance (no cuff weights weight wrapped around your thigh just above your kneecap), 4 = move the limb against some resistance (cuff weights weight wrapped around your thigh just above your kneecap) and 5 = normal motor strength against resistance. TUG is a performance test to measure functional mobility. The test requirements will be presented as the subject rises from a chair, walks 3.0 m easily to reach a mark placed on the floor, turns around at the 3.0 m mark, returns to the starting point and sits on the chair. The time the subject takes to complete the test is defined as the TUG score. Patients' movement with aid within 24 h will be encouraged when the motor strength was at least two. The postoperative patient satisfaction and incidence of adverse effects will be recorded. Patient satisfaction will be measured by a self administered satisfaction scale (very satisfied, somewhat satisfied, somewhat dissatisfied, very dissatisfied).

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to III.
2. Aged 40 to 70 years.
3. Both sexes.
4. Patients scheduled for unilateral total knee replacement.

Exclusion Criteria:

1. Patients with spinal malformation
2. Patients with liver impairment
3. Patients with renal impairment
4. Patients younger than 40 years or older than 70 years
5. Patients with hypersensitivity to one of the used drugs
6. Patients with neuromuscular disorders and
7. Coagulopathy disorders
8. Patients scheduled for revision knee arthroplasty or those who had a past history of previous surgery or trauma to the knee

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the total postoperative morphine consumption during the first two postoperative days. | 48 hours
  The primary outcome will be the total postoperative morphine consumption during the first two postoperative days.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abouseeda MM, Rashed MM, Hussein MM, Nady RF, Ehab AM. A Comparative Study Between Ultrasound-Guided Genicular Nerve Block Combined With Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee Block versus Adductor Canal Block in Total Knee Replacement. Anesthesiol Res Pract. 2025 May 22;2025:8937826. doi: 10.1155/anrp/8937826. eCollection 2025. PMID 40444065